CLINICAL TRIAL: NCT01935960
Title: A Randomized, Double-Blind, Phase I Dose-Escalation Study of the Novel Retinoid 9cUAB30
Brief Title: Retinoid 9cUAB30 in Preventing Cancer in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2013-01655; NCI-2013-01655 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UW13022 (Other: University of Wisconsin Chemoprevention Consortium); UWI10-16-01R (Other: DCP); N01CN35153 (NIH); P30CA014520 (NIH); NCT01999127 (obsolete NCT alias)
Record Dates: First submitted 2013-09-03; First posted 2013-09-05 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Healthy Subject
MeSH Terms: interventions — UAB 30

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (retinoid 9cUAB30) (Experimental): Participants receive retinoid 9cUAB30 PO QD on days 1 and 8-36. Treatment continues in the absence of unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Retinoid 9cUAB30
- Arm II (placebo) (Placebo Comparator): Participants receive a placebo PO QD on days 1 and 8-36.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Drug: Retinoid 9cUAB30 — Given PO
  Other Names: 9cUAB30
  Arms: Arm I (retinoid 9cUAB30)

SUMMARY:
This randomized phase I trial studies the side effects and best dose of retinoid 9cUAB30 in preventing cancer in healthy volunteers. The use of retinoid 9cUAB30 may keep cancer from forming in healthy volunteers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicities and recommended phase II dose of 9cUAB30 (retinoid 9cUAB30).

II. To characterize the urine and plasma single dose and steady state pharmacokinetics of 9cUAB30 in normal volunteers.

SECONDARY OBJECTIVES:

I. To correlate the pharmacokinetics of 9cUAB30 with toxicity. II. To compare observed toxicity between placebo controls and each dose level. III. To assess for any change in single dose pharmacokinetics (PK) after repeat dosing (day 1 vs. day 36).

OUTLINE: This is a dose-escalation study. Participants are randomized to 1 of 2 treatment arms.

ARM I: Participants receive retinoid 9cUAB30 orally (PO) once daily (QD) on days 1 and 8-36. Treatment continues in the absence of unacceptable toxicity.

ARM II: Participants receive a placebo PO QD on days 1 and 8-36.

After completion of study treatment, patients are followed up at 7 and 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Normal volunteers, either male or female
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 or Karnofsky >= 70%
* White blood cell (WBC) >= 3000/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin > 10 g/dL
* Bilirubin =< upper limit of institutional normal
* Aspartate aminotransferase (AST) =< upper limit of institutional normal
* Creatinine within institutional normal limits
* Sodium, potassium, chloride, bicarbonate: all =< upper limit of institutional normal
* Fasting triglycerides =< 1.5 x upper limit of normal (ULN)
* Fasting cholesterol =< 1.5 x ULN
* Participants must agree to discontinue all vitamin supplements while taking study medication and for thirty days past the last dose of study medication
* Heterosexual women and men must agree to use TWO effective forms of birth control for the duration of study participation and for 30 days following the last dose of study medication

  * Men must agree not to donate sperm during the study and for three months after receiving the last dose of study drug
  * The following persons are not considered to be able to father or bear children and therefore are eligible to participate without the use of concurrent birth control:

    * Female with bilateral oophorectomy and/or hysterectomy
    * Female with fallopian tubes cut, tied, or sealed
    * Female with sterilization implant (e.g. Adiana, Essure) placed > 3 months prior to randomization
    * Female post-menopausal (> 1 year since last menses)
    * Male with vasectomy > 3 months prior to randomization
  * One of the following methods of birth control must be used by women of childbearing potential:

    * Combined oral contraceptive pill in continuous use for > 30 days prior to study entry
    * Vaginal ring (e.g. NuvaRing) in continuous use for > 30 days prior to study entry
    * Skin patch (e.g. Ortho Evra) in continuous use for > 30 days prior to study entry
    * Injection (e.g. Depo-Provera, Noristerat) in continuous use for > 30 days prior to study entry
    * Copper intrauterine device (IUD) (e.g. ParaGard)
  * Note: The following hormonal methods are NOT acceptable:

    * Low dose progesterone only oral contraceptive pill ("mini pills" e.g. Micronor, Nor-Q.D., Ovrette)
    * Norplant subdermal implant
    * Mirena Hormonal Implanted Uterine Device (IUD)
  * In addition to the above method of contraception, one of the following methods of contraception will ALSO be used for the duration of study participation and for 30 days following the last dose of study medication:

    * Diaphragm, cervical cap, or cervical shield with spermicide
    * Contraceptive sponge (e.g. Today Sponge)
    * Condom (male or female type) plus spermicide
* Females of child-bearing potential must have a negative pregnancy test within the current menstrual cycle and within 7 days before starting drug
* Participants must have the ability to understand, and the willingness to sign, a written informed consent document

Exclusion Criteria:

* Participants may not be taking medications that might interact with 9cUAB30
* Participants may not be taking lipid lowering agents
* Participants may not receive any other investigational agents within 30 days of enrollment nor during study participation
* Participants with a history of allergic reactions attributed to compounds of similar chemical or biologic composition of retinoids
* Participants with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Breastfeeding must be discontinued for the duration of study participation and for one month after the last dose of the study agent if the mother is treated with 9cUAB30
* Individuals known to be human immunodeficiency virus (HIV)-positive may not participate in this study
* Individuals with a history of cancer diagnosis or reoccurrence < 5 years from study entry may not participate; however, individuals with a history of squamous or basal cell carcinoma of the skin < 5 years from study entry will not be excluded from this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of retinoid 9cUAB30, based on maximum tolerated dose (MTD), defined as the highest dose level with < 25% of treated patients experiencing a grade 2 toxicity or any treated patients experiencing a grade 3 or higher toxicity | Up to 30 days after completion of study treatment
  Graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Urine & plasma single dose & steady state PK of retinoid 9cUAB30, including maximum concentration (Cmax), time to peak concentration (Tmax), area under curve (AUC)0-least quantifiable concentration (lqc), AUC0-infinity, half-life (T½), and clearance (CL) | Baseline; 30, 45, 60, and 90 minutes; 2, 4, 6, 8, 12, 16, 20, and 24 hours on day 1; and 8, 15, 22, 29, 36, and 43 days
  Basic pharmacokinetic and summary pharmacokinetic measures from the extensive plasma sampling on days 1 and 36, and levels obtained from single plasma and urine samples taken on days 8, 15, 22, and 29 will be summarized with basic statistics, including means, standard errors, medians, and interquartile ranges by dose, visit, and time point, as available.

SECONDARY OUTCOMES:
Change in single dose pharmacokinetics, including Cmax, Tmax, AUC0-lqc, AUC0-infinity, T1/2, and CL | Day 1 to day 36
  The pharmacokinetics of retinoid 9cUAB30 will be compared between day 1 and day 36 using one-sample t-tests, or Wilcoxon signed-rank tests as appropriate in order to evaluate the single vs. steady state levels. An appropriate regression model will be used to explore the relationship of dose with change in PK: logarithmic transformations will be used as necessary.
Incidence of toxicity, graded according to the CTCAE version 4.0 | Up to 30 days after completion of study treatment
  Patient toxicity will be summarized by the presence or absence of any toxicities, worst CTCAE grade, and strongest investigator defined relationship will all be examined and characterized by dose. Correlations between the different PK measures of retinoid 9cUAB30 and the different measures of toxicity will be estimated with polyserial correlation. To compare toxicities at each dose level to placebo, the Chi-square test will be used for the presence or absence of toxicities, and Wilcoxon rank-sum tests will be used for CTCAE grade and investigator defined relationship data.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kolesar, Principal Investigator — University of Wisconsin Chemoprevention Consortium
Locations (3):
- United States (3):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin